CLINICAL TRIAL: NCT04599777
Title: Transcatheter Arterial Chemoembolization Combined With Sintilimab and Bevacizumab for Advanced Hepatocellular Carcinoma: An Open-label, Single-arm, Single-center, Prospective Study
Brief Title: TACE Combined With Sorafenib and Tislelizumab for Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-03
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma Non-resectable
MeSH Terms: interventions — Sorafenib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE-Sor-Tis (Experimental): TACE combined with sorafenib and tislelizumab.
  Interventions: Drug: TACE combined with sorafenib and tislelizumab

INTERVENTIONS:
Drug: TACE combined with sorafenib and tislelizumab — Sorafenib (400mg P.O. Bid) and tislelizumab (200mg I.V. q3w) will be started at 3-7 days after the first TACE. TACE will be repeated if clinically indicated. Treatment of tislelizumab will last up to 24 months. Patients will be allowed to have sorafenib or tislelizumab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

SUMMARY:
This study will evaluate the efficacy and safety of transcatheter arterial chemoembolization (TACE) combined with sorafenib and tislelizumab in patients with advanced hepatocellullar carcinoma (HCC).

DETAILED DESCRIPTION:
This is a Phase II study to evaluate the efficacy and safety of TACE combined with sorafenib and tislelizumab in patients with advanced HCC.

30 subjects with advanced HCC (Barcelona-Clinic- Liver-Cancer [BCLC] stage C, or China liver cancer staging [CNLC] IIIa and IIIb) will be enrolled in the study.

Both sorafenib (400mg P.O. Bid) and tislelizumab (200mg I.V. q3w) will be started at 3-7 days after the first TACE. TACE will be repeated if clinically indicated based on the evaluation of follow-up laboratory and imaging examination. Sorafenib will last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Sorafenib administration will be delayed in cases of grade ≥2 hand-foot syndrome, grade >3 hematologic toxicities or grade ≥3 hypertension. After recovery, sorafenib will be reintroduced at a reduced dose according the sorafenib dose delay and reduction guidelines. Treatment of tislelizumab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Patients will be allowed to have sorafenib or tislelizumab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Advanced HCC (BCLC stage C, or CNLC IIIa and IIIb ) with diagnosis confirmed by histology/cytology or clinically
* Disease not amenable to curative therapies but amenable to TACE
* At least one measurable untreated lesion
* No prior systemic therapy for HCC
* Child-Pugh score 5-7
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* Adequate organ and hematologic function
* Life expectancy of at least 3 months
* For women of childbearing potential and for men: agreement to remain abstinent

Exclusion Criteria:

* Diagnosis of fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Diffuse HCC
* Portal vein tumor thrombus (PVTT) involves the main trunk and contralateral branch or upper mesenteric vein
* Inferior vena cava tumor thrombus
* Metastatic disease that involves major airways or blood vessels
* Symptomatic, untreated or progressing central nervous system metastasis
* Uncontrolled tumor-related pain
* Patients who received prior systemic therapy, immunotherapy, TACE, transcatheter arterial radioembolization (TARE), transcatheter arterial embolization (TAE), hepatic arterial infusion chemotherapy (HAIC) or radiation therapy for HCC
* Treatment with systemic immunostimulatory agents
* Use of herbal therapies or traditional Chinese medicines with anti-cancer activity within 2 weeks
* History of malignancy other than HCC within 5 years prior to screening, except for malignancies with a negligible risk of metastasis or death
* Uncontrolled ascites, hydrothorax or pericardial effusion
* Prior esophageal and/or gastric varices bleeding within 6 months prior to initiation of study treatment
* Prior life-threatening blood loss or grade 3/4 gastrointestinal bleeding requiring blood infusion, endoscopic or surgical intervention within 3 months
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding
* History of gastrointestinal (GI) perforation and/or fistula in the past 6 months history of GI obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection, complicated by chronic diarrhea), Crohn's disease, ulcerative colitis or long-term chronic diarrhea
* History of hepatic encephalopathy
* History of organ and stem cell transplantation
* Long-term daily treatment with a non-steroidal anti-inflammatory drug (NSAID)
* Use of immunosuppressive drugs in the past 4 weeks, excluding the routes of topical glucocorticoids or physiological doses of systemic glucocorticoids (ie no more than 10 mg/day of prednisone or equivalent). Temporary use of glucocorticoids for dyspnea symptoms such as asthma and chronic obstructive pulmonary disease is allowed
* History of idiopathic pulmonary fibrosis, interstitial pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* Active tuberculosis
* Active severe infection; use of antibiotics within 2 weeks prior to injection of tislelizumab
* Autoimmune disease or immune deficiency
* Inadequately controlled hypertension; history of hypertensive crisis or hypertensive encephalopathy
* Bleeding diathesis or significant coagulopathy
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture underwent major surgery (craniotomy, thoracotomy or open surgery) within 4 weeks; non-recovery from side effects of these procedure
* History of venous thromboembolism in the past 6 months, but implantable IV ports or catheter-derived thrombosis, superficial venous thrombosis, or thrombosis after conventional anticoagulant therapy are excluded
* Current or recent use of aspirin or treatment with dipyramidole, ticlopidine, clopidogrel, or cilostazol uncontrolled metabolic disorder, non-malignant organ or systemic disease or secondary carcinomatous reaction, with high medical risk and/or uncertainty of life expectancy evaluation
* Other acute or chronic diseases, mental illness, or abnormal laboratory test results that may lead to the following outcomes: increase the risk of participating in study or study drug administration, or interfere with the interpretation of the study results and considered by investigator as "NOT" eligible to participate in this study
* Female patients who are pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 24 months
  The time from initiation of treatment until the date of death from any cause.

SECONDARY OUTCOMES:
Adverse Events (AEs) | 24 months
  Number of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), AE of special interest (AESI), serious adverse event (SAE), assessed by NCI CTCAE v5.0.
Progression free survival (PFS) assessed by investigators according to Response Evalutaion Criteria in Solid Tumors (RECIST) v1.1 and immune-related RECIST (irRECIST). | 24 months
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.
Objective response rate (ORR) assessed by investigators according to RECIST 1.1 and irRECIST. | 24 months
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR).
Disease control rate (DCR) assessed by investigators according to RECIST 1.1 and irRECIST. | 24 months
  The percentage of patients who had a tumor response rating of CR, PR, or stable disease (SD).
Duration of response (DOR) assessed by investigators according to RECIST 1.1 and irRECIST. | 24 months
  The time from the first occurrence of a documented objective response to disease progression (PD) or death.
PFS assessed by investigators according to Modified RECIST (mRECIST). | 24 months
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.
ORR assessed by investigators according to mRECIST. | 24 months
  The percentage of patients who had a best overall tumor response rating of CR or PR.
DCR assessed by investigators according to mRECIST. | 24 months
  The percentage of patients who had a tumor response rating of CR, PR, or SD.
DOR assessed by investigators according to mRECIST. | 24 months
  The time from the first occurrence of a documented objective response to PD or death.

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, Dr., Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - The 2nd Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong